CLINICAL TRIAL: NCT03067142
Title: "Pilot Study: Proteomics of Primary Hyperoxaluria Type 1 (PH1): A Rare Calcium Oxalate Stone Disease"
Brief Title: Proteomics of Primary Hyperoxaluria Type 1
Acronym: PH1
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Mayo Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 6409; 2U54DK083908-06 (NIH)
Record Dates: First submitted 2017-02-09; First posted 2017-03-01 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Primary Hyperoxaluria Type 1
MeSH Terms: conditions — Primary hyperoxaluria type 1 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 (Phase 1): PH1: Cross-Sectional/Observational
  Interventions: Other: Observational
- Cohort 2 (Phase 1): Controls: Cross-Sectional/Observational
  Interventions: Other: Observational
- Cohort 3 (Phase 2): PH1: Longitudinal/Observational
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Not an interventional study. Analyses of previously collected urine specimens and data on estimated kidney filtering function.

SUMMARY:
The purpose of this study is to identify unique urine protein markers of Primary Hyperoxaluria type 1 (PH1) compared to healthy controls. Urine protein markers can be identified by "proteomic" analyses in which proteins are processed in a lab to break them down into smaller building blocks. Using analytical chemistry techniques and specialized equipment many proteins can be identified and measured. Most proteins are found in healthy living cells while subtle changes in these proteins or the presence of different markers reflect abnormal processes and patterns of disease. When identified in disease, protein biomarkers can help to determine if a disease responds to new types of therapies. In this study, changes in urine proteomic patterns over time, their association with change in estimated (calculated) kidney filtering function, and the relative risk for progression of PH1 will be determined. Additionally, as part of the study, the investigators will measure urinary proteins and peptides that are markers of kidney tissue protection (for healthy healing of the kidneys from ongoing damage from high urine oxalate levels, oxalate crystals and stones) to establish if and when these markers are prospectively decreased in PH1 urine. Longitudinal studies of urine "proteomics" may assist in identifying the mechanisms behind PH1-related progression of kidney failure and might contribute important information towards future identification and development of effective therapies to slow or prevent kidney failure in PH1.

DETAILED DESCRIPTION:
Primary hyperoxaluria type 1 (PH1) is a rare genetically inherited disorder seen in 1:100,000-150,000 people and is often underdiagnosed in children. PH1 is characterized by abnormally high levels of oxalate in the blood and urine, crystals in the urine, frequent formation of kidney stones, and hardening (calcification) of the kidneys called "nephrocalcinosis." Identification and evaluation of proteins and peptides (biomarkers) in the urine of PH1 patients may provide insight into the process of kidney damage that occurs over time in PH1 by evaluating these markers at some point after diagnosis and over long-term. By studying biomarker patterns in the urine of PH1 patients that are collected over the course of their disease, information about changes in biomarker patterns over time may provide important clues about those patients at a higher risk for faster progression to end stage kidney failure and may serve as important outcomes for new therapies in the future, too.

Primary study objective: Identify the unique urine proteomic markers of PH1 versus healthy intra-familial sibling controls of PHI patient specimens at one point in time (cross-sectionally).

Secondary study objective: Determine change over time in urine proteomic patterns, their association with change in estimated (calculated) kidney filtering function, and the relative risk for progression of PH1 and kidney disease progression.

Tertiary study objective: Establish if and when, in the course of PH1, the protective effects of the body (and kidneys) for normal kidney tissue healing are decreased/ lost as evidenced by the long-term change in biomarker patterns.

The primary endpoints of this study include standard clinical endpoints (data that a kidney doctor would look at as a PH1 patient would be followed over time in the clinic), as they best reflect PH1 disease progression: (a) estimated glomerular filtration rate (eGFR), known as kidney filtering function; (b) urine oxalate; and (c) plasma oxalate (when eGFR < 40 ml/min/1.73 m2, which is when kidney function is significantly decreased).

The goal of the Rare Kidney Stone Consortium (RKSC) is to advance understanding and treatment of severe, rare forms of nephrolithiasis that cause marked excretion of insoluble minerals important in stone formation in which patients experience recurring stones from childhood onward and are at risk for chronic kidney disease. End state renal disease is common in PH1. Importantly, these conditions are rare enough that there has been minimal sharing of information and expertise among clinicians and scientists, a situation that has slowed progress toward effective treatments. Over the last 6 years, RKSC has formed secure, web-based registries and tissue banks open for collaborative projects.

About this Study: This is a pilot investigation using previously collected and archived (1) cross-sectional 24 hr. urine samples from PH1 patients (n=20) and healthy sibling controls (n=18) and (2) longitudinally collected 24 hr. urine samples from patients with PH1 enrolled in the RKSC registry bank (n=55). No new samples will be collected.

Additional information that will be collected (or provided with the urine specimens) as part of this study: De-identified data from each patient's health history, medications and supplements taken; history of kidney stones (and their chemical make-up); gender, current age, height, weight; old measurements of urine acidity, and blood oxalate, urine oxalate, calcium, citrate, and creatinine (from muscle breakdown) concentrations, and urine super saturation.

ELIGIBILITY:
Inclusion Criteria:

* Have a previously collected 24 hour urine sample from the Mayo Clinic's Rare Kidney Stone Consortium (RKSC) biobank or previously stored at Lurie Children's Hospital (Chicago, IL), a portion of which has been archived (frozen) for future research because you are a patient who has been diagnosed with Primary Hyperoxaluria type 1 (PH1) that is documented by one of the following: (1) PH1 mutation confirmed and/or (2) liver biopsy confirmed; OR
* Have a previously collected 24 hour urine sample, a portion of which has been archived (frozen) for future research, because you are a healthy sibling of a PH1 patient, as described above.

Exclusion Criteria:

* Have a previously collected 24 hour urine sample because you are a hyperoxaluric patient due to other causes (including secondary hyperoxaluria);
* Have PH1 and have had a 24 hour sample collected but a portion of that specimen has not been archived (frozen) for future research;
* Do not have PH1.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients with Primary Hyperoxaluria Type 1 (PH1) OR
  2. Healthy siblings of those PH1 patients (to serve as "controls)
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Phase 1: Urine proteomic markers. | Baseline
  (1) Quantitative Mass Spectrometry analyses will be completed on previously collected, de-identified, and archived urine specimens (collected at only one time point) from patients with Primary Hyperoxaluria type 1 (PH1) and from healthy controls to determine unique protein markers in the urine of PH1 patients, taking into account archived data collected about: (a) known genetic PH1 mutations; (b) concomitant estimated kidney filtering function; (c) urine and plasma oxalate concentrations (using the measure of plasma oxalate when kidney function is low) (d) the level of kidney function (called a "stage"); and (e) any medications and supplements & their dose and frequency taken for differences in disease (PH1) versus a healthy state. To accomplish this, urine specimens and data which were previously collected, de-identified, and archived will be provided by Mayo Clinic (Rochester, MN) and Ann & Robert H. Lurie Children's Hospital of Chicago (Chicago, IL).

SECONDARY OUTCOMES:
Phase 2: Urine proteomic marker patterns and their change over time related to progression of chronic kidney disease in primary hyperoxaluria type 1 (PH1). | 5 years
  Quantitative Mass Spectrometry analyses of previously collected, archived, and de-identified serial urine specimens (collected in up to/more than 5 years of follow-up) from patients with Primary Hyperoxaluria type 1 (PH1) will be completed to determine if a change occurs in: (1) urine proteomic patterns (proteins and peptides) over time using previously collected data on: (a) estimated kidney filtering function declines (indicating kidney disease progression) and (b) oxalate concentrations in the urine (or plasma) continue to rise. Statistical analyses will determine the relationship between the urine protein/peptide pattern changes over time to kidney disease progression in PH1. All previously collected, de-identified, and archived data and urine specimens will be provided by Mayo Clinic (Rochester, MN).
Phase 2: Establish by urine proteome pattern changes if & when normal healing processes of the kidneys are lost, which reflect progressive kidney damage. | 5 years
  Establish if and when, in the 5 year serial follow-up of Primary Hyperoxaluria type 1 (PH1) urine specimens, normal kidney tissue healing is decreased/lost (down regulated) and pathologic kidney tissue damage increases (upregulated). This will be evidenced by the long-term change in biomarker patterns and progressive loss of kidney filtering function. This will be accomplished using: (1) standard identification of specific urine protein and peptides using known databases and (2) statistical analyses for urine protein/peptide marker pattern development reflective of kidney pro-injury and irreversible kidney cell damage. (All serially collected, de-identified, and archived urine specimens and data will have been provided by Mayo Clinic, Rochester, MN).

CONTACTS AND LOCATIONS:
Overall Officials: Craig B Langman, MD, Principal Investigator — Ann & Robert H Lurie hildren's Hospital of Chicago, Division of Kidney Diseases

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lapolla A, Seraglia R, Molin L, Williams K, Cosma C, Reitano R, Sechi A, Ragazzi E, Traldi P. Low molecular weight proteins in urines from healthy subjects as well as diabetic, nephropathic and diabetic-nephropathic patients: a MALDI study. J Mass Spectrom. 2009 Mar;44(3):419-25. doi: 10.1002/jms.1520. PMID 19165811
- [Background] Metzger J, Kirsch T, Schiffer E, Ulger P, Mentes E, Brand K, Weissinger EM, Haubitz M, Mischak H, Herget-Rosenthal S. Urinary excretion of twenty peptides forms an early and accurate diagnostic pattern of acute kidney injury. Kidney Int. 2010 Dec;78(12):1252-62. doi: 10.1038/ki.2010.322. Epub 2010 Sep 8. PMID 20827258
- [Background] Kistler AD, Serra AL, Siwy J, Poster D, Krauer F, Torres VE, Mrug M, Grantham JJ, Bae KT, Bost JE, Mullen W, Wuthrich RP, Mischak H, Chapman AB. Urinary proteomic biomarkers for diagnosis and risk stratification of autosomal dominant polycystic kidney disease: a multicentric study. PLoS One. 2013;8(1):e53016. doi: 10.1371/journal.pone.0053016. Epub 2013 Jan 10. PMID 23326375
- [Background] Evan AP, Coe FL, Lingeman JE, Shao Y, Sommer AJ, Bledsoe SB, Anderson JC, Worcester EM. Mechanism of formation of human calcium oxalate renal stones on Randall's plaque. Anat Rec (Hoboken). 2007 Oct;290(10):1315-23. doi: 10.1002/ar.20580. PMID 17724713
- [Background] Yasui T, Fujita K, Hayashi Y, Ueda K, Kon S, Maeda M, Uede T, Kohri K. Quantification of osteopontin in the urine of healthy and stone-forming men. Urol Res. 1999 Aug;27(4):225-30. doi: 10.1007/s002400050114. PMID 10460890
- [Background] Zhang Y, Wen Z, Washburn MP, Florens L. Refinements to label free proteome quantitation: how to deal with peptides shared by multiple proteins. Anal Chem. 2010 Mar 15;82(6):2272-81. doi: 10.1021/ac9023999. PMID 20166708
- [Background] Pieper R. Preparation of urine samples for proteomic analysis. Methods Mol Biol. 2008;425:89-99. doi: 10.1007/978-1-60327-210-0_8. PMID 18369889
- [Background] McIlwain S, Mathews M, Bereman MS, Rubel EW, MacCoss MJ, Noble WS. Estimating relative abundances of proteins from shotgun proteomics data. BMC Bioinformatics. 2012 Nov 19;13:308. doi: 10.1186/1471-2105-13-308. PMID 23164367
- [Background] Skates SJ, Gillette MA, LaBaer J, Carr SA, Anderson L, Liebler DC, Ransohoff D, Rifai N, Kondratovich M, Tezak Z, Mansfield E, Oberg AL, Wright I, Barnes G, Gail M, Mesri M, Kinsinger CR, Rodriguez H, Boja ES. Statistical design for biospecimen cohort size in proteomics-based biomarker discovery and verification studies. J Proteome Res. 2013 Dec 6;12(12):5383-94. doi: 10.1021/pr400132j. Epub 2013 Oct 28. PMID 24063748